CLINICAL TRIAL: NCT05611008
Title: Seniors Empowered Via Big Data to Joint-manage Their Medication-related Risk of Falling in Primary Care
Brief Title: Testing the SNOWDROP Intervention: Using a Clinical Decision Support System and Patient Portal for Falls Prevention Among Older Patients in Primary Care
Acronym: SNOWDROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Responsible Party: Principal Investigator, Julia van Weert, Prof. dr. Julia van Weert, University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-PC-15274
Record Dates: First submitted 2022-10-18; First posted 2022-11-09 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Fall; Fall Injury; Fall Patients; Accidental Fall; Deprescribing
MeSH Terms: interventions — Patient Portals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention condition (Experimental)
  Interventions: Device: CDSS; Device: Patient Portal
- Control condition (No Intervention)

INTERVENTIONS:
Device: CDSS — A Clinical Decision Support System (CDSS) that calculates older patients' personalized fall risk and provides the GP with advice on how to adjust the patient's medication in order to lower the fall risk.
  Arms: Intervention condition
Device: Patient Portal — A patient portal that provides general information on falls and fall risk to the older patients and helps the patient to prepare for the consultation by filling out a Question Prompt List (QPL). The QPL is a list of possibly relevant questions and topics from which the patient can select those that are important to him/her. These will already be sent to the GP before the consultation takes place.
  Arms: Intervention condition

SUMMARY:
Falls are a leading cause of injuries among older patients. Medication use is a major risk factor for falls. Because we lack tools to assess individualized risks, general practitioners (GPs) struggle with fall-related medication management for older patients. Furthermore, these older patients are often not properly equipped to engage in the joint management of their medication. A Clinical Decision Support System (CDSS) for GPs and a patient portal for older patients may stimulate shared decision making between GPs and older patients when discussing the medication-related fall risk. The CDSS provides the GP with advice on how to alter medication in such a way that the fall risk decreases, and the patient portal helps the older patient to prepare for a consultation and to engage in the joint management of their medication.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* High fall risk
* Takes at least 1 Fall Risk Increasing Drug (FRID)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Shared decision making | During consultation
  This concerns the extent to which shared decision making between patient and GP during the consultation. This will be assessed using the Observer OPTION Multiple Chronic Conditions (OPTION-MCC). Consultation are audiotaped and will be coded on shared decision making using this coding scheme.

SECONDARY OUTCOMES:
Technology Acceptance Model (TAM; patient portal) | At baseline & two weeks after consultation
  The Technology Acceptance Model (TAM) measures the adoption of a new technology/system based on user attitudes in relation to the patient portal.
Website Satisfaction Scale (WSS; patient portal) | At baseline & two weeks after consultation
  The Website Satisfaction Scale (WSS) measures satisfaction with comprehensibility, satisfaction with attractiveness, and satisfaction with emotional support, in relation to the patient portal.
Patient portal usage | At baseline & two weeks after consultation
  Patients are asked if they used the patient portal and which components they used.
Beliefs About Medicines Questionnaire (BMQ) | Baseline & two weeks after consultation
  The Beliefs about Medicines Questionnaire measures beliefs about the necessity of medication and concerns about medication.
Netherlands Patient Information Recall Questionnaire (NPIRQ) | Two weeks after consultation
  The Netherlands Patient Information Recall Questionnaire consists of open questions measuring patients' recall of what was discussed and decided during the consultation.
Decisional Conflict Scale (DCS) | Two weeks after consultation
  The decisional conflict scale measures decisional conflict after the consultation related to five subscales: feeling informed, uncertainty, values clarity, support, and effective decision making.
Changes in medication | Baseline & two weeks after the consultation
  Changes in prescriptions of the medication as reported in the electronic health record.
Technology Acceptance Model (TAM; CDSS) | After the first consultation (study beginning) and after the last consultation (study completion after +/- 7 months)
  The Technology Acceptance Model (TAM) measures the adoption of a new technology/system based on user attitudes in relation to the CDSS to be answered by the GP. This is assessed by measuring Perceived Usefulness, Perceived Ease of Use, and Intention to use.
The Website Satisfaction Scale (WSS; CDSS) | After the first consultation (study beginning) and after the last consultation (study completion after +/- 7 months)
  The Website Satisfaction Scale (WSS) measures satisfaction with comprehensibility, satisfaction with attractiveness, and satisfaction with emotional support, in relation to the CDSS to be answered by the GP.
Evaluation of the consultation | Immediately after each consultation
  Four items to assess the consultation to be answered by the GP. The items assess to what extent the patient was representative, their opinion on the communication during the consultation, the extent to which they are satisfied with any decisions made and the difficulty of the consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Julia C.M. van Weert, Principal Investigator — Amsterdam School for Communication Research (ASCoR), University of Amsterdam
Locations (1):
- Huisartsenpraktijken, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Currently no plan